CLINICAL TRIAL: NCT04550611
Title: Efficacy of Mini-pool Intravenous Immunoglobulin (MP-IVIG) Prepared by Assiut University Hospital Blood Bank in Guillain-Barré Syndrome
Brief Title: Mini-pool Intravenous Immunoglobulin (MP-IVIG) in Guillain-Barré Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Ahmed Hassan Moubark, clinical pathology specialist at assiut university hospitals blood banks, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Guillain-Barré syndrome
Record Dates: First submitted 2020-08-27; First posted 2020-09-16 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-09

CONDITIONS: Guillain-Barre Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — Plasma Exchange; Plasmapheresis

STUDY DESIGN:
Intervention Model Description: The process of MP-IVIG preparation will involve the use of caprylic acid for purification and virus inactivation of Igs from mini-pools of 20 plasma donations collected in our Central blood transfusions( CBTS) in Assiut University Hospital (AUH). The equipment used for the process comprised disposable blood bags, hemodialyzers, and purification and microbial filters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini-pool Intravenous Immunoglobulin (MP-IVIG) (Experimental): will receive blood group -specific MP-IVIG in a regimen of 2 g/kg bodyweight, usually as 0.4 g/kg bodyweight per day for five consecutive days within two weak of onset of symptoms.
  Interventions: Other: Mini-pool Intravenous Immunoglobulin (MP-IVIG)
- plasmapheresis (Experimental): plasma exchange (plasmapheresis ) in a regimen of removing of 1.3 plasma volumes in each cycle for total of five cycle for five consecutive days within four weeks of onset of symptoms.
  Interventions: Other: plasma exchange

INTERVENTIONS:
Other: Mini-pool Intravenous Immunoglobulin (MP-IVIG) — The process of MP-IVIG preparation will involve the use of caprylic acid for purification and virus inactivation of Igs from mini-pools of 20 plasma donations collected in our CBTS in AUH. The equipment used for the process comprised disposable blood bags, hemodialyzers, and purification and microbial filters.
  Arms: Mini-pool Intravenous Immunoglobulin (MP-IVIG)
Other: plasma exchange — plasma exchange (plasmapheresis ) in a regimen of removing of 1.3 plasma volumes in each cycle for total of five cycle for five consecutive days within four weeks of onset of symptoms.
  Other Names: plasmapheresis
  Arms: plasmapheresis

SUMMARY:
1. study the pharmacokinetics of mini-pooled intravenous immunoglobulin( MP-IVIG)
2. to determine the efﬁcacy of intravenous immunoglobulin (IVIg) in hastening recovery and reducing the complications of Guillain-Barré syndrome (GBS).

   * The MP-IVIG was tolerated and presented no safety issues in a previous study and we will be confirmed by monitoring any adverse events (anaphylaxis and haemolysis) ( no or mild or moderate) and reporting them to ethical committee safety monitoring group.
   * Efficacy will be confirmed by:

     1. Patient able to walk
     2. Improvement of general health.
     3. Integration in to social live
3. to compare the efﬁcacy of IVIg to plasma exchange (PE) in hastening recovery and improving the condition of GBS

DETAILED DESCRIPTION:
Guillain-Barré syndrome (GBS) is a frequent cause of neuromuscular paralysis occurring at all ages. The incidence of GBS is reported to be 1.2-2.3 per 100,000 per year .

GBS is a post infectious disorder. The most frequently identified preceding infection is Campylobacter jejuni. Others are cytomegalovirus, Epstein-Barr virus, Mycoplasma pneumoniae, and Haemophilus influenzae . Many reports have documented the occurrence of GBS shortly after vaccinations, operations, or stressful events, but the causality and pathophysiology are still debated .

Rapidly progressive weakness is the core clinical feature of GBS. By definition, maximal weakness is reached within 4 weeks, but most patients reach it within 2 to 3 weeks. Thereafter, patients enter a plateau phase that ranges from days to several weeks or months . This phase is followed by a usually much slower and variable recovery phase. In Europe, about one-third of GBS patients remain able to walk ("mild patients") .about 25% of the GBS patients who are unable to walk ("severe patients") need artificial ventilation. This is predominantly due to weakness of the respiratory muscles. GBS has a great impact on social life and the ability to perform activities of daily life. therefore, GBS remains a severe disease for which better treatments are required .

. Magdy EL-Ekiaby, et al 2010 introduce the concept of small-scale ("minipool") plasma processing methods. The preparation of the Immunoglobulin G (IgG) plasma fractionation from 20 blood donations which are tested for anti-A and anti-B titre < 32. Implementable with minimum infrastructural requirements. They developed viral inactivation and protein purification technologies in single-use equipment to prepare virally safe solvent/detergent-filtered (S/D-F) plasma Producing a 90%pure immunoglobulin fraction in disposable single-use devices for transfusion .

IVIG adverse events (AEs) are not frequent; hemolysis after IVIG is a known, rare complication. Higher doses and non-O blood group are key risk factors. The incidence of post-IVIG hemolysis is estimated at 1 per 1000 IVIG treatment episodes, most of which occur within 2 days of exposure. Although the preparation of blood group specific IVIGs in industry is a complex issue because of the pooling of thousands of plasma donations per batch, the preparation of blood group-specific mini-pool IVIG (MP-IVIG) is possible because each pool consists of only 20 plasma donations. Blood group-matched MP-IVIG is assumed to reduce the incidence of IVIG-associated hemolysis, which is largely caused by the presence of anti-A and anti-B agglutinins reacting with non-O blood group recipients.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 18-40 years.
* Both sex are include
* The study will include patient diagnosed as Guillain-Barré syndrome (mild) cases in neuropsychiatric hospital at Assiut university hospitals.

Exclusion Criteria:

* • Patient has severe form of Guillain-Barré syndrome (GBS) according to GBS disability score

  * Patient with renal impairment
  * Patient with hepatic cell failure

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy ofMini-pool Intravenous Immunoglobulin (MP-IVIG) assessed by patients achieve score more than or equal 2 according to GBS disability score | 6 MONTHS
  Guillain-Barré syndrome disability scale Score Description 0 A healthy state
  1. Minor symptoms and capable of running
  2. Able to walk 10m or more without assistance but unable to run
  3. Able to walk 10m across an open space with help
  4. Bedridden or chairbound
  5. Requiring assisted ventilation for at least part of the day
  6. Dead
Safety of MP-IVIG assessed by percentage of adverse Events: Overall percentage of adverse events | 72 hour after adminstration of MP-IVIG and between infusions period
  Overall percentage of adverse events as hemolysis and anaphylaxis headache and other complains that occur during 72 hours of following an infusion of MP-IVIG will be assessed by1) vital sign(pulse,blood pressure,Respiratory rate and temperature 2)Hemolysis by hemoglobin level, Lactate dehydrogenase( LDH),bilirubin level.2)between infusions by home diaries.
Study the pharmacokinetics- MP-IVIG trough levels | predose sample
  MP-IVIG trough level concentration values of serum total IgG pre the MP-IVIG infusion (if applicable).
Study the pharmacokinetics MP-IVIG plasma concentration -time curve [ | (1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days) post-dose ]
  Blood samples for analysis of pharmacokinetics MP-IVIG plasma concentration -time curve were obtained and analysed Blood samples for analysis of pharmacokinetics MP-IVIG plasma concentration -time curve were obtained and analysed
Study the pharmacokinetics MP-IVIG half-life | (1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days) post-dose ]
  Blood samples for analysis of pharmacokinetics MP-IVIG haf-life were obtained and analysed
Study the pharmacokinetics MP-IVIG area under the curve | (1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days) post-dose ]
  Blood samples for analysis of pharmacokinetics MP-IVIG haf-life were obtained and analysed
Study the pharmacokinetics MP-IVIG Cmax | (1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days) post-dose ]
  Blood samples for analysis of pharmacokinetics MP-IVIG Cmax were obtained and analysed
Study the pharmacokinetics of MP-IVIG-Tmax. | (1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days) post-dose ]
  Blood samples for analysis of pharmacokinetics MP-IVIG Tmax were obtained and analysed
Study the pharmacokinetics of MP-IVIG elimination rate constant(s). : ( | 1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days) post-dose ]
  Blood samples for analysis of pharmacokinetics MP-IVIG elimination rate constant(s) were obtained and analysed

SECONDARY OUTCOMES:
• compare the efﬁcacy of IVIg to plasma exchange (PE) according to GBS disability score | 6 MONTHS
  Guillain-Barré syndrome disability scale Score Description 0 A healthy state
  1. Minor symptoms and capable of running
  2. Able to walk 10m or more without assistance but unable to run
  3. Able to walk 10m across an open space with help
  4. Bedridden or chairbound
  5. Requiring assisted ventilation for at least part of the day
  6. Dead

CONTACTS AND LOCATIONS:
Overall Officials: Maha A Mohamed, Prof, Study Director — Assiut University

REFERENCES:
- [Background] van Doorn PA, Ruts L, Jacobs BC. Clinical features, pathogenesis, and treatment of Guillain-Barre syndrome. Lancet Neurol. 2008 Oct;7(10):939-50. doi: 10.1016/S1474-4422(08)70215-1. PMID 18848313
- [Background] El-Ekiaby M, Vargas M, Sayed M, Gorgy G, Goubran H, Radosevic M, Burnouf T. Minipool caprylic acid fractionation of plasma using disposable equipment: a practical method to enhance immunoglobulin supply in developing countries. PLoS Negl Trop Dis. 2015 Feb 26;9(2):e0003501. doi: 10.1371/journal.pntd.0003501. eCollection 2015 Feb. PMID 25719558
- [Background] El-Ekiaby M, Sayed MA, Caron C, Burnouf S, El-Sharkawy N, Goubran H, Radosevich M, Goudemand J, Blum D, de Melo L, Soulie V, Adam J, Burnouf T. Solvent-detergent filtered (S/D-F) fresh frozen plasma and cryoprecipitate minipools prepared in a newly designed integral disposable processing bag system. Transfus Med. 2010 Feb;20(1):48-61. doi: 10.1111/j.1365-3148.2009.00963.x. Epub 2009 Sep 23. PMID 19778318
- [Background] Winiecki S, Baer B, Chege W, Jankosky C, Mintz P, Baker M, Woodworth T, Nguyen M. Complementary use of passive surveillance and Mini-Sentinel to better characterize hemolysis after immune globulin. Transfusion. 2015 Jul;55 Suppl 2:S28-35. doi: 10.1111/trf.13116. PMID 26174895
- [Background] Ojha R, Karn R(2019):Clinical outcome of intravenous immunoglobulin in the treatment of Guillain Barre Syndrome in a Nepalese tertiary centre. Nep Med J 2019;2(1):133-7.
- [Result] Hughes RA, Cornblath DR. Guillain-Barre syndrome. Lancet. 2005 Nov 5;366(9497):1653-66. doi: 10.1016/S0140-6736(05)67665-9. PMID 16271648